CLINICAL TRIAL: NCT00158002
Title: An Open-Label Study of Topiramate in Pediatric Subjects With Basilar/Hemiplegic Migraine
Brief Title: A Study of Topiramate in Pediatric Subjects With Basilar/Hemiplegic Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Monarch Medical Research (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: CAPSS 299
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Basilar Migraine
Keywords: Basilar/Hemiplegic Migraine; Prophylaxis
MeSH Terms: conditions — Migraine with Aura | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The objective of this study is to assess the long-term safety and effectiveness of topiramate in the prevention of basilar and hemiplegic migraine in children and adolescents.

DETAILED DESCRIPTION:
This is a single-center, open-label study consisting of 3 phases: Blinded Transition Phase, Open-Label Maintenance Phase, and Taper/Exit Phase. Subjects who have either succesfully completed the CAPSS-271 protocol or who discontinued the CAPSS-271 study due to lack of effectiveness after completing at least 2 weeks of maintenance treatment will be eligible to enroll.

ELIGIBILITY:
Inclusion Criteria:

* Must have either completed the Double-Blind Phase of CAPSS-271 or discontinued the Double-Blind Phase of CAPSS-271 due to lack of efficacy after a minimum of 2 weeks of maintenance treatment.
* Must continue to meet the specific inclusion criteria outlined in CAPSS-271.
* Female subjects must be premenarchal, surgically sterile (hysterectomy, tubal ligation or otherwise incapable of pregnancy); or practicing an effective method of birth control (e.g., intrauterine device, double-barrier method, male partner sterilization) at study entry and throughout the study; or hormonal contraceptives for at least a 3-month period prior to the start of the study and throughout the study, or be practicing abstinence and agree to continue abstinence or to use an acceptable method of contraception (as listed above) should sexual activity commence. In addition, female subjects of childbearing potential must have a negative urine pregnancy test at Open-Label Visit 1 (Day 1).
* Must be able to read and comprehend written instructions and be willing to complete all headache records and questionnaires as required by the protocol.
* After full explanation of the study, subjects, or their parent/legally authorized representative(s), must demonstrate their willingness to participate by signing an informed consent form. If applicable, pediatric subjects capable of giving assent must sign the assent form.

Exclusion Criteria:

* Subjects who have developed a more painful condition than their headache pain.
* Subjects taking any of the prohibited concomitant medications (See Concomitant Medications section).
* Subjects who are pregnant.
* Subjects with liver function tests ³ 2 times the upper limit of the normal range.
* In the investigator's opinion, subjects with poor compliance during the CAPSS-271 study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2004-02; Study Completion 2006-08

PRIMARY OUTCOMES:
Reduction of average monthly migraine days
Reduction in frequency, severity and duration of basilar or hemiplegic aura symptoms
Reduction in migraine pain severity and duration
Migraine episode and headache episode frequency
Total headache days
Proportion of responders (i.e., the proportion of subjects who experience a 50% reduction in migraine-days and migraine episodes)

SECONDARY OUTCOMES:
Cumulative frequency of migraine days and migraine episodes
Use of acute/abortive medications
Migraine episode and headache episode frequency
Total headache days
Migraine-associated symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Lewis, MD, Principal Investigator — Monarch Medical Research
Locations (1):
- Monarch Medical Research - Child and Adolescent Neurology, Norfolk, Virginia, United States